CLINICAL TRIAL: NCT04304937
Title: Validation of a Swedish Version of a Short Patient-Reported-Outcome-Measure for Superficial Venous Insufficiency
Brief Title: Validation of Swedish Short PROM för Venous Insufficiency
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Skandinaviska Forskningsstiftelsen för Åderbråck och andra Vensjukdomar (Unknown)
Responsible Party: Principal Investigator, Karolina Hultman, MD PhD, Karolinska Institutet
Other Study IDs: 2017/1824 - 31/2
Record Dates: First submitted 2020-03-09; First posted 2020-03-12 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Superficial Venous Insufficiency; Quality of Life; Change After Treatment
Keywords: Patient reported outcome measure
MeSH Terms: interventions — Patient Reported Outcome Measures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: test-retest at baseline and 7 days later
  Interventions: Other: patient reported outcome measure
- Cohort 2: test at baseline and 8 weeks post treatment
  Interventions: Other: patient reported outcome measure

INTERVENTIONS:
Other: patient reported outcome measure — 2 questionnaires are tested against each other

SUMMARY:
Validation of a new short Swedish patient reported outcome measure for superficial venous insufficiency. Analysis of its capacity to measure quality of life and its responsiveness to change caused by treatment.

ELIGIBILITY:
Inclusion Criteria:

* agrees to participate, diagnosed with superficial venous insufficiency C2-C6

Exclusion Criteria:

* does not want to participate, less than C2, does not submit the answered questionnaires

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: consecutive patients at chosen clinics diagnosed with superficial venous insufficiency C2-C6
Sampling Method: Non-Probability Sample
Enrollment: 257 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
the short PROM is valid for measurement of quality of life and detects change caused by treatment | baseline and 8 weeks

CONTACTS AND LOCATIONS:
Locations (3):
- Sweden (3):
  - Karlskoga venöst centrum, Karlskoga
  - Åderbråckscentrum, Malmo
  - Narvakliniken Åderbråck, Stockholm

IPD SHARING:
Plan to Share IPD: Undecided